CLINICAL TRIAL: NCT06408831
Title: The Effect of Web-Based Cyber Sexual Violence Training and Consultancy on Cyber Sexual Violence Experience, Sensitivity and Cyber Security
Brief Title: The Effect of Web-Based Cyber Sexual Violence Training on Cyber Sexual Violence Experience, Sensitivity and Security
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sehadet, specialist nurse, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IU-SBE-ST-01
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Cyberbullying
Keywords: cyber; sexuality; web; education; consultancy
MeSH Terms: conditions — Cyberbullying; Sexuality

STUDY DESIGN:
Intervention Model Description: two groups with control group without training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classroom Teaching University Students Intervention Group (Active Comparator): A special username and password will be given to the intervention group, which is randomly assigned to the female students of the classroom teaching department, to log in to the website, and they will be given a special access to the website. Afterwards, training on cyber sexual violence will be given within the scope of the literature. The scales will be applied to the students again after 12 weeks in order to see the effect of the behavior.
  Interventions: Behavioral: Classroom Teaching University Students Intervention Group
- Kindergarten Teaching University Students Control Group (No Intervention): Participant Introduction Form, Cyber Sexual Violence Scale, Sensitivity Scale for Cyber Bullying (SZBÖ) Young Adult Form, Ensuring Personal Cyber Security Scale will be applied to the control group of kindergarten teaching female students as a pre-test. The Participant Introduction Form, Cyber Sexual Violence Scale, Sensitivity Scale for Cyber Bullying (SZSS) Young Adult Form, and Ensuring Personal Cyber Security Scale will be applied to the control group again after an average of 8-10 weeks without any intervention. In accordance with ethical principles, after the final results of the control group are collected, the videos in the training content will be sent to the control group.

INTERVENTIONS:
Behavioral: Classroom Teaching University Students Intervention Group — Web-based cyber sexual violence training and counseling will be provided to female classroom teaching students, who are the intervention group, and the effect of the intervention on cyber sexual violence experience, sensitivity and cyber security will be examined.
  Arms: Classroom Teaching University Students Intervention Group

SUMMARY:
The aim of this study is to provide web-based cyber sexual violence training with a model (Knowledge, Motivation, Behavior Skills (IMB) Model) to female university students, who are one of the groups that are vulnerable to being victimized in terms of cyber sexual violence.

DETAILED DESCRIPTION:
This research was conducted with a pre-test-post-test control group trial model to measure the effect of web-based cyber sexual violence training and counseling based on the information-motivation-behavioral skills (IMB) model given to young people on cyber sexual violence experience, sensitivity and cyber security ensuring behavior. It was planned as a study. The sample of our research will consist of female students from the Department of Primary Education and Kindergarten Teaching at Harran University. The sample size of the study was calculated with Z test logistic regression using the G*Power 3.1.9.2 program, taking the gender risk of sexual cyberbullying as a reference in Klein and Cooper's study. According to the power analysis, it was calculated that the sample of the research should have at least 85 people in the groups with an effect size of 0.20 and a 95% confidence interval determined by a 5% error level, with a 995% representative power of the universe. It was planned to include an equal number of students from the first, second, third and fourth grades of the Primary School Teaching and Kindergarten Teaching departments in the research using the stratified sampling method. Considering the losses from each group, it was planned to select a total of 200 people from the experimental (100 female classroom teaching students) and control group (100 female kindergarten teaching students). Criteria for inclusion in the research; not being medically diagnosed with a psychological disease, being between the ages of 18-26, being single, being a classroom or kindergarten teacher student, using a smartphone, and having the opportunity to access the internet on a daily basis; Exclusion criteria were determined as failure to complete the intervention and failure to fill out the data collection form. Research data will be obtained using the Participant Introduction Form, the Sensitivity Scale on Cyberbullying (SZSS) Young Adult Form, and the Personal Cybersecurity Ensuring Scale. Data will be collected via online interview method on the web. After the forms are applied to the experimental and control groups, the experimental group will be given a username and password to access the established website and they will receive the prepared training in video and word format. It will be checked whether the students in the experimental group have watched the educational videos, reminder messages will be sent and calls will be made to them to watch all uploaded educational videos. After training and counseling, the same tests will be applied again to the experimental group. For the control group, only pre-test and post-test will be administered without any intervention. Descriptive statistics such as percentage, arithmetic mean (X) and standard deviation (SD) were used to examine the socio-demographic characteristics of the students. Chi-square test, paired sample t-test, independent samples t-test were used to determine whether there was a difference between the control variables and the experimental and control groups. -test, Bonferroni test will be used to determine which group the difference between the groups originates from, independent samples t-test will be used to determine whether there is a difference between the mean scores of the scales in the experimental and control groups, and paired sample t-test will be used to compare the mean scores of the pre-test and post-test. With the results obtained from this study, the effect of web-based cyber sexual violence training and counseling given to university students on cyber sexual violence victimization, sensitivity to cyber bullying and ensuring cyber security will be determined. In the literature review, no studies were found on web-based training and consultancy against cyber sexual violence. As a result of the data obtained from this study, it is thought that the cyber sensitivity and security of the web-based training and consultancy to be given to university students against cyber sexual violence can be determined and valuable data can be provided for the use of relevant professionals.

ELIGIBILITY:
Inclusion Criteria:

* Not being medically diagnosed with a psychological disease
* Being between the ages of 18-26
* Being single
* Being a classroom and kindergarten teaching student
* Using a smartphone
* Having the opportunity to access the internet on a daily basis

Exclusion Criteria:

* Inability to complete the intervention
* Not filling out the data collection form

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Studies have stated that cyber sexual violence may be predominantly related to gender and sexuality, and that young women are more likely to be victims than men.
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Cyber Sexual Violence Scale | 6 months
  The scale assessing sexual violence experienced online consists of 18 items. The scale is a five-point Likert type (always = 5, often = 4, sometimes = 3, rarely = 2, never = 1). The lowest score that can be obtained from the scale is 18 and the highest score is 90. The scale consists of two subscales: "Unwanted sexual texts" and "Unwanted sexual desire". In the Turkish validity and reliability study of the scale, Cronbach Alpha value was found to be 0.94 for the total score of the scale, 0.94 for the Sexual texts sub-dimension and 0.90 for the Unwanted sexual desire sub-dimension.
Sensitivity Scale on Cyberbullying Young Adult Form | 6 months
  The scale is scored on a three-point scale as No (1), Sometimes (2), Yes (3). The scale is one-dimensional and gives scores between 7 and 21. A high score indicates high sensitivity. Since the scale has not been normed, there is no cut-off score. Cronbach's alpha coefficients were calculated for both versions to see how reducing the number of scales affected the internal consistency of the scale. "While the alpha value for the 13-item version was .87, the value for the seven-item version was 0.83, and it was found that there was a minimal decrease in internal consistency after reducing it to six items."
Ensuring Personal Cyber Security Scale | 6 months
  The scale consists of 5 factors and 25 items. These factors are named as "protecting personal privacy" (10 items), "avoiding the untrustworthy" (4 items), "taking precautions" (5 items), "protecting payment information" (2 items) and "leaving no trace" (4 items). . The Cronbach Alpha reliability coefficient of the 5-point Likert type scale was calculated as 0.735. The reliability coefficients for the sub-dimensions are "protecting personal privacy" 0.763, "avoiding the untrustworthy" 0.771, "taking precautions" 0.704, "protecting payment information" 0.829 and "leaving no trace" 0.557. The scale is suitable for individuals aged 18 and over.

IPD SHARING:
Plan to Share IPD: No